CLINICAL TRIAL: NCT04457453
Title: Comparison of Direct Laryngoscope and Video Laryngoscope During Endotracheal Intubation in Sellick and Trendelenburg Position to Prevent Pulmonary Aspiration
Brief Title: Comparison of Direct and Video Laryngoscope During Endotracheal Intubation in Sellick and Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AJIRB-MED-OBS-19-507
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Intubation;Difficult
Keywords: Trendelenburg position; Sellick position; pulmonary aspiration; video laryngoscope
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): intubation with direct laryngoscope in sniffing position
  Interventions: Other: Macintosh in sniffing position
- direct laryngoscope in Trendelenburg and Sellick position (Experimental): intubation with direct laryngoscope in Trendelenburg and Sellick position
  Interventions: Other: Macintosh in Trendelenburg position and Sellick position
- video laryngoscope in Trendelenburg and Sellick position (Experimental): intubation with video laryngoscope in Trendelenburg and Sellick position
  Interventions: Other: AceScope in Trendelenburg position and Sellick position

INTERVENTIONS:
Other: Macintosh in sniffing position — Macintosh direct intubation in sniffing position
  Arms: control group
Other: Macintosh in Trendelenburg position and Sellick position — Macintosh direct laryngoscopic intubation in Trendelenburg position and Sellick position
  Arms: direct laryngoscope in Trendelenburg and Sellick position
Other: AceScope in Trendelenburg position and Sellick position — AceScope videolaryngoscopic intubation in Trendelenburg position and Sellick position
  Arms: video laryngoscope in Trendelenburg and Sellick position

SUMMARY:
Pulmonary aspiration during tracheal intubation for anesthesia can cause fatal respiratory complications. Takenaka's study of mannequins reported that the risk of airway contamination by reflux gastric contents could be minimized by applying a 15-degree Trendelenburg position and a Sellick position with neck extention. However, the clinical performance of tracheal intubation in this position has not been studied. Also, the difference between the effects of direct laryngoscope and video laryngoscope on tracheal intubation is not known yet.

Therefore, this study aims to compare the intubation time among intubation through direct laryngoscope and video laryngoscope in the Sellick and Trendelenburg position, and intubation in the conventional sniffing position.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 19 years old
* ASA I or II
* Patients who need nasotracheal intubation for surgery

Exclusion Criteria:

* Anatomical deformity in head and neck
* Patients who have risk of pulmonary aspiration
* Patients with cervical deformities or pain
* BMI >35

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Intubation time | within 5 minutes
  from endotracheal tube pass the teeth to end-tidal CO2 appear

SECONDARY OUTCOMES:
Intubation difficulty score | within 5 minutes
  Intubation difficulty scale (IDS) score

CONTACTS AND LOCATIONS:
Overall Officials: yun jeong chae, Ph.D, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou universitiy school of medicine, Suwon, Gyeong-gi Do, South Korea